CLINICAL TRIAL: NCT00489255
Title: A Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of Trimethobenzamide (Tigan®) in the Control of Nausea and Vomiting During Initiation and Continued Treatment With Subcutaneous Apomorphine (Apokyn®) in Apomorphine-naïve Subjects With Parkinson's Disease Suffering From Acute Intermittent "Off" Episodes, With Phased Withdrawal of Subjects From Tigan® to Placebo
Brief Title: Safety/Efficacy of Tigan® to Control Nausea/Vomiting Experienced During Apokyn® Initiation and Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Collaborators: INC Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-47-52844-003; APO-4PD-01
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Anti-emetic; Nausea; Vomiting
MeSH Terms: conditions — Parkinson Disease; Nausea; Vomiting | interventions — trimethobenzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trimethobenzamide (Tigan®) (Experimental)
  Interventions: Drug: Tigan®
- Inactive substance (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tigan® — Oral capsule, 300mg three times daily
  Arms: Trimethobenzamide (Tigan®)
Drug: Placebo — Oral capsule, three times daily
  Arms: Inactive substance

SUMMARY:
The purposes of the study are to determine:

i. To assess the efficacy of Tigan® (trimethobenzamide) in preventing nausea and vomiting when initiating therapy with Apokyn® (apomorphine)

ii. To determine the optimal duration for continuation of Tigan® following initiation of Apokyn® therapy

iii. To assess the safety of Tigan® in combination with Apokyn®

iv. To characterize the pharmacokinetic (PK) profile of apomorphine in subjects treated concomitantly with and without Tigan®

DETAILED DESCRIPTION:
Initial randomization is Tigan or Placebo (3:1) with phased withdrawal of Tigan to Placebo after 4 and 8 weeks. Subjects completing 4 weeks Tigan re-randomized to Tigan or Placebo (2:1) with patients completing 8 weeks Tigan re-randomized to receive Tigan or Placebo (1:1). Subjects randomized to Placebo over the previous 4 weeks assigned to continue on Placebo for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or over
* Subjects with advanced Parkinson's disease with disabling hypomobility ("off" episodes) who are to be initiated with Apokyn® by intermittent subcutaneous injection
* Able to swallow Tigan®/placebo capsules
* Subjects willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
* Women of child bearing potential must have a negative serum pregnancy test (beta hCG) prior to receiving study drug and must be using an appropriate form of contraception
* Willing and able to provide informed consent

Exclusion Criteria:

* Hypersensitive to apomorphine hydrochloride or any of the ingredients of Apokyn® (notably sodium metabisulfite)
* Hypersensitive to trimethobenzamide or any of the ingredients of Tigan®
* Previous treatment with Apokyn®
* Participation in any other clinical trial within 14 days of the present trial
* Contraindications to Apokyn® or Tigan®
* Currently taking, or likely to need to take at any time during the course of the study, any 5HT3 antagonist (ondansetron, alosetron, granisetron, palonosetron or dolasetron)
* Malignant melanoma or a history of previously treated malignant melanoma
* Pregnancy or breast feeding
* Receipt of any investigational (i.e. unapproved) medication within 30 days of starting the present trial
* Any significant medical disorder, condition, concomitant medication or psychiatric disorder according to DSM-IV criteria which would, in the opinion of the investigator, represent a hazard to the subject or prevent the subject from completing the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (27):
- United States (27):
  - Barrow Neurological Movement Disorder Clinic, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Coastal Neurological Medical Group Inc., La Jolla, California
  - Neurosearch, Inc., Reseda, California
  - Neurosearch II, Inc., Ventura, California
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Neurology at Shands Medical Center, Gainesville, Florida
  - University of Florida at Jacksonville, Jacksonville, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Charlotte Neurological Services, Port Charlotte, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - USF Parkinson's Disease and Movement Disorders Center of Excellence, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - NorthShore University Health System, Glenview, Illinois
  - Iowa Health Physicians, Des Moines, Iowa
  - Parkinson's & Movements Disorders Center of Maryland, Elkridge, Maryland
  - Quest Research Institute, Bingham Farms, Michigan
  - Henry Ford Health System - Franklin Point, Southfield, Michigan
  - Parkinson's Disease and Movement Disorders Center of Long Island, Commack, New York
  - Kingston Neurological Associates, Kingston, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Neurological Institute, Cleveland Clinic, Cleveland, Ohio
  - Neurology Specialist of Dallas P.A, Dallas, Texas
  - Parkinson's Disease and Movement Disorders Center, Baylor College of Medicine, Houston, Texas
  - Neurology Associates, P.A., San Antonio, Texas
  - East Texas Medical Center, Tyler, Texas
  - Sentara Neurological Associates, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 24 investigational sites in the United States (US).
Pre-assignment Details: Number of participants "STARTED" does not match "Enrollment, Actual" (in protocol section) due to re-randomization design of the study & phased withdrawal of subjects from Tigan to placebo. Some subjects were included on one treatment in one period and re-randomized to a different treatment in a later period.
Groups:
- Trimethobenzamide (Tigan®): Tigan® : Oral capsule, 300mg three times daily.
- Tigan:Placebo: Placebo : Oral capsule, three times daily.
Period: Screening and Initial Randomization
Arm/Group | Trimethobenzamide (Tigan®) | Tigan:Placebo
Started | 145 (Total randomized subjects to receive Tigan) | 49 (Total randomized subjects to receive placebo)
Completed | 136 | 46
Not Completed | 9 | 3
Not completed — Discontinued prior to taking study drug | 9 | 3
Period: Period 1: Days 1 to 28
Arm/Group | Trimethobenzamide (Tigan®) | Tigan:Placebo
Started | 136 | 46
Completed and Follow Period 2 | 94 | 29
Completed But Discontinued Study | 13 | 5
Completed | 107 | 34
Not Completed | 29 | 12
Not completed — Adverse Event | 21 | 8
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Physician Decision | 1 | 4
Not completed — Noncompliance | 2 | 0
Period: Period 2: Days 29 to 56
Arm/Group | Trimethobenzamide (Tigan®) | Tigan:Placebo
Started | 64 | 59 (Re-randomized participants is 26.Sample sizes differed due to withdrawal&re-randomization design.)
Completed and Follow Period 3 | 58 | 52 (Re-randomized participants is 26.Sample sizes differed due to withdrawal&re-randomization design.)
Completed But Discontinued Study | 3 | 3 (Re-randomized participants is 2.Sample sizes differed due to withdrawal&re-randomization design.)
Completed | 61 | 55 (Re-randomized participants is 26.Sample sizes differed due to withdrawal&re-randomization design.)
Not Completed | 3 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 0 | 3
Period: Period 3: Days 57 to 84
Arm/Group | Trimethobenzamide (Tigan®) | Tigan:Placebo
Started | 28 | 82 (Re-randomized participants is 30.Sample sizes differed due to withdrawal&re-randomization design.)
Completed | 24 | 78 (Re-randomized participants is 27.Sample sizes differed due to withdrawal&re-randomization design.)
Not Completed | 4 | 4
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo : Oral capsule, three times daily.
- Total: Total of all reporting groups
Arm/Group | Trimethobenzamide (Tigan®) | Placebo | Total
Number analyzed (Participants) | 134 | 46 | 180
Age, Continuous [Median (Full Range); unit: years] — Period 1:
  Overall Number of Baseline Participants in 'Trimethobenzamide (Tigan®)' arm is 134.
  Overall Number of Baseline Participants in 'Placebo' arm is 46.
  years | 65.5 [24.0 to 93.0] | 63.5 [49.0 to 79.0] | 65.0 [24.0 to 93.0]
Age, Continuous [Median (Full Range); unit: years] — Period 2 (Re-randomized patients):
  Overall Number of Baseline Participants in 'Trimethobenzamide (Tigan®)' arm is 64.
  Overall Number of Baseline Participants in 'Placebo' arm is 30 (re-randomized) and 59 (all placebo).
  years | 64.0 [33.0 to 86.0] | 65.5 [24.0 to 85.0] | 64.0 [24.0 to 86.0]
Age, Continuous [Median (Full Range); unit: years] — Period 3 (Re-randomized patients):
  Overall Number of Baseline Participants in 'Trimethobenzamide (Tigan®)' arm is 28.
  Overall Number of Baseline Participants in 'Placebo' arm is is 30 (re-randomized) and 82 (all placebo).
  years | 66.5 [41.0 to 86.0] | 63.0 [33 to 84.0] | 64.0 [24.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants] — Data for Period 1.
  Period 2 & 3 are as follows:
  Period 2, Re-randomized patients
  Female: 19 participants in 'Trimethobenzamide (Tigan®)' arm and 11 participants in 'Placebo' arm.
  Male: 45 participants in 'Trimethobenzamide (Tigan®)' arm and 19 participants in 'Placebo' arm.
  Period 3, Re-randomized patients
  Female: 7 participants in 'Trimethobenzamide (Tigan®)' arm and 8 participants in 'Placebo' arm.
  Male: 21 participants in 'Trimethobenzamide (Tigan®)' arm and 22 participants in 'Placebo' arm.
  Participants
    Female | 42 | 13 | 55
    Male | 92 | 33 | 125
Unified Parkinson's Disease Rating Scale (UPDRS) total score for Period 1 [Mean (Standard Deviation); unit: Score on a scale] — The UPDRS is a 4-part rating tool to follow the longitudinal course of Parkinson's disease. The four sections in the scale are 1. Mentation, Behavior and Mood, 2. Activities of Daily Living (ADL), 3. Motor Exam and 4. Complications of Therapy. UPDRS total score range from 0 to 199, with 199 indicative of the worst and 0 no disability.
  Score on a scale | 49.2 (21.26) | 47.8 (17.83) | 48.8 (20.40)
UPDRS motor score for Period 1 [Mean (Standard Deviation); unit: Score on a scale] — Part III (Motor Examination) of the UPDRS contains 14 items designed to assess the severity of the cardinal motor findings (e.g., tremor, rigidity, bradykinesia, postural instability, etc.) in patients with Parkinson's disease. UPDRS motor score range from 0 to 56, with 56 indicative of the worst and 0 no disability.
  Score on a scale | 25.7 (15.07) | 25.2 (12.25) | 25.6 (14.37)
UPDRS total score for Period 2 [Mean (Standard Deviation); unit: Score on a scale] — The UPDRS is a 4-part rating tool to follow the longitudinal course of Parkinson's disease. The four sections in the scale are 1. Mentation, Behavior and Mood, 2. Activities of Daily Living (ADL), 3. Motor Exam and 4. Complications of Therapy. UPDRS total score range from 0 to 199, with 199 indicative of the worst and 0 no disability.
  Score on a scale | 46.7 (21.32) | 47.6 (18.83) | 47.1 (20.09)
UPDRS motor score for Period 2 [Mean (Standard Deviation); unit: Score on a scale] — Part III (Motor Examination) of the UPDRS contains 14 items designed to assess the severity of the cardinal motor findings (e.g., tremor, rigidity, bradykinesia, postural instability, etc.) in patients with Parkinson's disease. UPDRS motor score range from 0 to 56, with 56 indicative of the worst and 0 no disability.
  Score on a scale | 24.3 (15.50) | 25.5 (12.60) | 24.9 (14.14)
UPDRS total score for Period 3 [Mean (Standard Deviation); unit: Score on a scale] — The UPDRS is a 4-part rating tool to follow the longitudinal course of Parkinson's disease. The four sections in the scale are 1. Mentation, Behavior and Mood, 2. Activities of Daily Living (ADL), 3. Motor Exam and 4. Complications of Therapy. UPDRS total score range from 0 to 199, with 199 indicative of the worst and 0 no disability.
  Score on a scale | 48.1 (17.84) | 47.5 (20.87) | 47.6 (20.06)
UPDRS motor score for Period 3 [Mean (Standard Deviation); unit: Score on a scale] — Part III (Motor Examination) of the UPDRS contains 14 items designed to assess the severity of the cardinal motor findings (e.g., tremor, rigidity, bradykinesia, postural instability, etc.) in patients with Parkinson's disease. UPDRS motor score range from 0 to 56, with 56 indicative of the worst and 0 no disability.
  Score on a scale | 25.5 (13.58) | 25.1 (14.69) | 25.2 (14.35)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Nausea and/or Vomiting During the Initial Titration of Apokyn® at the Visit on Day 1
Time Frame: Day 1 (Period 1, Visit 2)
Population: Primary efficacy analyses performed on the Intention-to-Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 130 | 44
participants
  Subjects who experienced nausea &/or vomiting[Yes] | 21 [0.17 to 1.11] | 10 [0.17 to 1.11]
  Subjects who experienced nausea &/or vomiting [No] | 109 | 34
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; The null hypothesis was no difference between treatments; Test type: Superiority or Other; p = 0.09, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test for treatment was stratified by site; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.17 to 1.11]

2. Secondary Outcome: Incidence of Nausea and/or Vomiting for Period 1
Time Frame: Days 1-28
Population: Secondary efficacy analyses performed on the Intention-to-Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 130 | 44
participants
  Yes | 48 | 24
  No | 82 | 20
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.21 to 0.90]

3. Secondary Outcome: Incidence of Nausea and/or Vomiting for Period 2
Time Frame: Days 29-56
Population: Secondary efficacy analyses performed on the Intention-to-Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 63 | 30
participants
  Yes | 15 | 14
  No | 48 | 16
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.25, 95% CI 2-sided [0.09 to 0.70]

4. Secondary Outcome: Incidence of Nausea and/or Vomiting for Period 3
Time Frame: Days 57-84
Population: Secondary efficacy analyses performed on the Intention-to-Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 27 | 30
participants
  Yes | 9 | 10
  No | 18 | 20
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.65, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.23 to 2.48]

5. Secondary Outcome: Modified Index of Nausea, Vomiting and Retching (INVR) Scores - Total Experience Score for Period 1
Description: The INVR is an 8-item, 5 point Likert-type measurement of the patient's perceived experience of nausea, vomiting and retching. Modified INVR scores collected once daily, rather than twice a day. INVR total score range from 0 to 32, with 32 indicative of the worst and 0 no symptom.
Time Frame: Days 1-28
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 130 | 44
score on a scale | 0.51 (1.504) | 0.80 (1.755)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.32, ANOVA; Treatment effect in ANOVA was adjusted for site; Median Difference (Net) = -0.21, 95% CI 2-sided [-0.64 to 0.21]

6. Secondary Outcome: Modified Index of Nausea, Vomiting and Retching (INVR) Scores - Total Experience Score for Period 2
Description: as for outcome 5
Time Frame: Days 29-56
Population: Secondary efficacy analyses performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 63 | 30
score on a scale | 0.19 (0.491) | 1.27 (2.568)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.001, ANOVA; Median Difference (Net) = -1.07, 95% CI 2-sided [-1.71 to -0.43]

7. Secondary Outcome: Modified Index of Nausea, Vomiting and Retching (INVR) Scores - Total Experience Score for Period 3
Description: as for outcome 5
Time Frame: Days 57-84
Population: Secondary efficacy analyses performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 27 | 30
score on a scale | 0.27 (0.684) | 0.21 (0.392)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.95, ANOVA; Median Difference (Net) = -0.01, 95% CI 2-sided [-0.20 to 0.19]

8. Secondary Outcome: Subject Global Evaluation of Randomized Study Medication for Period 1
Description: The subject global evaluation of Tigan/placebo was completed by the subject at the visits in response to the question "Overall, how would you rate the study medication you received for nausea/vomiting?" Response choices were excellent, very good, good, fair, or poor.
Time Frame: Day 28 (Visit 3)
Population: This secondary efficacy analysis was performed on the total number of subjects who responded to the evaluation within the Intention-to-Treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 107 | 34
participants
  Excellent | 61 | 20
  Very good | 23 | 5
  Good | 10 | 3
  Fair | 6 | 3
  Poor | 7 | 3
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.88, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test (row mean score) with rigid scores, stratified by site

9. Secondary Outcome: Subject Global Evaluation of Randomized Study Medication for Period 2
Description: as for outcome 8
Time Frame: Day 56 (Visit 4)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 61 | 29
participants
  Excellent | 38 | 15
  Very good | 16 | 4
  Good | 2 | 2
  Fair | 3 | 2
  Poor | 2 | 6
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.019, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test (row mean score) with rigid scores, stratified by site

10. Secondary Outcome: Subject Global Evaluation of Randomized Study Medication for Period 3
Description: as for outcome 8
Time Frame: Day 84 (Visit 5)
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 26 | 29
participants
  Excellent | 17 | 24
  Very good | 4 | 2
  Good | 3 | 0
  Fair | 0 | 0
  Poor | 2 | 3
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.29, Cochran-Mantel-Haenszel

11. Secondary Outcome: Median Time to 'on' for Visit 2/Period 1 Injection 1
Description: Time to "on" (relief of immobility) was measured 20 minutes after administration of Apokyn and before discharge at the clinic; calculated as the difference between the recorded time of "on" and time of injection.
Time Frame: Day 1 (Visit 2)
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 130 | 44
minutes | 25.0 [16.0 to 31.0] | 20.0 [14.0 to 34.0]
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.17, Regression, Cox — Cox's proportional hazards model with site and treatment (Tigan/placebo) as factors; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.5 to 1.1]

12. Secondary Outcome: Median Time to 'on' for Visit 2/Period 1 Injection 2
Description: as for outcome 11
Time Frame: Day 1 (Visit 2)
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 47 | 10
minutes | 20.0 [15.0 to 36.0] | 16.5 [6.0 to 20.0]
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.008, Regression, Cox — Cox's proportional hazards model with site and treatment (Tigan/placebo) as factors; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.1 to 0.7]

13. Secondary Outcome: Median Time to 'on' for Visit 3/End of Period 1 Injection
Description: as for outcome 11
Time Frame: Day 28
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 94 | 31
minutes | 12.0 [10.0 to 15.0] | 10.0 [8.0 to 11.0]
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.49, Regression, Cox — Cox's proportional hazards model with site and treatment (Tigan/placebo) as factors; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.6 to 1.3]

14. Secondary Outcome: Median Time to 'on' for Visit 4/End of Period 2 Injection
Description: as for outcome 11
Time Frame: Day 56 (Visit 4)
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 59 | 27
minutes | 10.0 [10.0 to 13.0] | 12.0 [10.0 to 15.0]
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.4, Regression, Cox; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.7 to 2.1]

15. Secondary Outcome: Median Time to 'on' for Visit 5/End of Period 3 Injection
Description: as for outcome 11
Time Frame: Day 84 (Visit 5)
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 24 | 27
minutes | 10.0 [9.0 to 15.0] | 10.0 [10.0 to 15.0]
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.62, Regression, Cox — Cox's proportional hazards model with site and treatment (Tigan/placebo) as factors; Hazard Ratio (HR) = 1.2, 95% CI [0.6 to 2.3]

16. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 (Motor Section) for Visit 2, Pre Apokyn Dose, Period 1
Description: Part 3 (Motor Examination) of the UPDRS contains 14 items designed to assess the severity of the cardinal motor findings (e.g., tremor, rigidity, bradykinesia, postural instability, etc.) in patients with Parkinson's disease. UPDRS motor score range from 0 to 56, with 56 indicative of the worst and 0 no disability.
Time Frame: Day 1 (Visit 2)
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 130 | 44
score on a scale | 35.5 (13.72) | 35.3 (13.31)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.96, ANOVA; ANCOVA model with baseline score (score at Visit 1/Screening) as a covariate, and site and treatment as factors; Mean Difference (Net) = 0.08, 95% CI 2-sided [-3.59 to 3.76]

17. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 (Motor Section) for Visit 3, Pre Apokyn Dose, Period 1
Description: as for outcome 16
Time Frame: Day 28
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 106 | 33
score on a scale | 34.0 (14.27) | 34.2 (13.08)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.93, ANOVA; Mean Difference (Net) = -0.18, 95% CI 2-sided [-4.37 to 4.02]

18. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 (Motor Section) for Visit 3, Post Apokyn Dose, Period 1
Description: as for outcome 16
Time Frame: Day 28
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 94 | 30
score on a scale | 20.8 (13.21) | 21.1 (12.94)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.84, ANOVA; Mean Difference (Net) = 0.39, 95% CI 2-sided [-4.12 to 3.34]

19. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 (Motor Section) for Visit 4, Pre Apokyn Dose, Period 2
Description: as for outcome 16
Time Frame: Day 56 (Visit 4)
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 60 | 27
score on a scale | 37.1 (15.07) | 33.3 (11.19)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.25, ANOVA; Mean Difference (Net) = 2.97, 95% CI 2-sided [-2.17 to 8.11]

20. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 (Motor Section) for Visit 4, Post Apokyn Dose, Period 2
Description: as for outcome 16
Time Frame: Day 56 (Visit 4)
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 59 | 27
score on a scale | 20.9 (12.86) | 19.0 (7.01)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.46, ANOVA; Mean Difference (Net) = 1.47, 95% CI 2-sided [-2.47 to 5.40]

21. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 (Motor Section) for Visit 5, Pre Apokyn Dose, Period 3
Description: as for outcome 16
Time Frame: Day 84 (Visit 5)
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 26 | 28
score on a scale | 37.7 (13.42) | 34.3 (14.95)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.33, ANOVA; Mean Difference (Net) = 2.96, 95% CI 2-sided [-3.13 to 9.06]

22. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 (Motor Section) for Visit 5, Post Apokyn Dose, Period 3
Description: as for outcome 16
Time Frame: Day 56 (Visit 4)
Population: This secondary efficacy analysis was performed on the Intention-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Number analyzed (Participants) | 24 | 27
score on a scale | 22.6 (13.52) | 21.4 (14.87)
Statistical Analysis 1: Comparison: Trimethobenzamide (Tigan®) vs Placebo; Test type: Superiority or Other; p = 0.93, ANOVA; Mean Difference (Net) = 0.27, 95% CI 2-sided [-5.57 to 6.11]

ADVERSE EVENTS:
Arm/Group | Trimethobenzamide (Tigan®) | Placebo
Serious Adverse Events (participants affected / at risk) | 4/134 | 6/106
Other Adverse Events (participants affected / at risk) | 86/134 | 57/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trimethobenzamide (Tigan®) (N=134) | Placebo (N=106)
Dysphagia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Chest pain (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trimethobenzamide (Tigan®) (N=134) | Placebo (N=106)
Somnolence (Nervous system disorders) | 26 | 14
Dizziness (Nervous system disorders) | 19 | 11
Dyskinesia (Nervous system disorders) | 14 | 8
Headache (Nervous system disorders) | 11 | 2
Yawning (Respiratory, thoracic and mediastinal disorders) | 19 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Fall (Injury, poisoning and procedural complications) | 10 | 1
Fatigue (General disorders) | 6 | 3
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No